CLINICAL TRIAL: NCT07398599
Title: To Explore the Efficacy and Safety of Double-dose Third-generation EGFR-TKI Combined With Bevacizumab and Intrathecal Chemotherapy in Advanced NSCLC Patients With Progressive Leptomeningeal Metastasis After Prior Standard-dose Third-generation EGFR-TKI Treatment.
Brief Title: Double-Dose Third-Generation EGFR-TKI Plus Bevacizumab and Intrathecal Chemotherapy for Refractory Leptomeningeal Metastatic NSCLC: A Phase II Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2025-640
Record Dates: First submitted 2026-01-29; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Leptomeningeal Metastasis; Lung Neoplasms, Non-Small Cell Lung Cancer
Keywords: Leptomeningeal Metastasis; non-small cell lung cancer
MeSH Terms: conditions — Meningeal Carcinomatosis; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- a combined regimen consisting of double-dose third-generation EGFR-TKI, bevacizumab, and intrathecal (Experimental)
  Interventions: Combination Product: a combined regimen consisting of double-dose third-generation EGFR-TKI, bevacizumab, and intrathecal chemotherapy in patients

INTERVENTIONS:
Combination Product: a combined regimen consisting of double-dose third-generation EGFR-TKI, bevacizumab, and intrathecal chemotherapy in patients — The combined treatment includes three components: double-dose third-generation EGFR-TKI (oral osimertinib 160mg once daily, furmonertinib 160mg once daily, or almonertinib 220mg once daily); intrathecal pemetrexed (administered via lumbar puncture, Ommaya reservoir, or intrathecal pump, with induction phase: 10mg twice weekly for 4 weeks, maintenance phase: 10mg once weekly for 4 weeks, consolidation phase: 30mg every 4 weeks until disease progression or intolerable toxicity); and bevacizumab 7.5mg/kg administered intravenously.

SUMMARY:
The goal of this clinical trial is to explore the efficacy and safety of double-dose third-generation EGFR-TKI combined with bevacizumab and intrathecal chemotherapy in treating advanced non-small cell lung cancer (NSCLC) patients with leptomeningeal metastasis that progressed after prior standard-dose third-generation EGFR-TKI treatment. It also aims to investigate the correlation between cerebrospinal fluid genetic characteristics and prognosis as well as subsequent efficacy prediction in patients with leptomeningeal metastasis after resistance to standard-dose third-generation EGFR-TKI. The main questions it intends to answer are:

Does this combined treatment regimen improve leptomeningeal metastasis response rate (LM-ORR) evaluated by RANO-LM? What adverse events occur in patients during the treatment with this combined regimen? Researchers will conduct a single-arm phase II prospective study to assess the effectiveness and safety of the combined treatment, without a control group comparison.

Participants will:

Receive double-dose third-generation EGFR-TKI (osimertinib 160mg qd, furmonertinib 160mg qd, or almonertinib 220mg qd) + intrathecal pemetrexed (induction phase: 10mg twice a week for 4 weeks; maintenance phase: 10mg once a week for 4 weeks; consolidation phase: 30mg every 4 weeks until disease progression or intolerable toxicity) + bevacizumab 7.5mg/kg.

Undergo screening assessments within 28 days before enrollment, including tumor imaging, laboratory tests, and cerebrospinal fluid examination.

During the treatment period, conduct regular checkups and tests (such as blood routine, blood biochemistry, electrocardiogram, and imaging examinations) according to the protocol (once every 4 weeks in the first two treatment cycles, then once every 8 weeks).

Complete quality of life assessment using the QLQ-C30 scale every 4 weeks and record changes in neurological symptoms and ECOG scores.

DETAILED DESCRIPTION:
1. Study Overview This is a prospective, single-arm Phase II interventional clinical trial initiated by the Second Affiliated Hospital of Nanchang University, with funding from the Wu Jieping Medical Foundation. The study will be conducted from December 2025 to December 2027 (Version V1.0, dated November 20, 2025) and led by Principal Investigator Cai Jing (contact number: 0791-86260752). The core objective is to evaluate the efficacy and safety of a combined regimen consisting of double-dose third-generation EGFR-TKI, bevacizumab, and intrathecal chemotherapy in patients with advanced non-small cell lung cancer (NSCLC) who have developed leptomeningeal metastasis (LM) after prior standard-dose third-generation EGFR-TKI treatment. Additionally, the study explores the correlation between cerebrospinal fluid (CSF) genetic characteristics and prognosis, as well as predictive value for subsequent efficacy, in patients with LM following resistance to standard-dose third-generation EGFR-TKI.
2. Study Population 2.1 Inclusion Criteria Participants must meet all the following criteria to be enrolled: aged ≥18 years at the time of signing the informed consent form, regardless of gender; histologically or cytologically confirmed advanced or metastatic NSCLC, staged as IV according to the 8th edition of the IASLC TNM classification (2015); presence of EGFR-sensitive mutations (exon 19 deletion or exon 21 mutation), with LM progression after prior standard-dose third-generation EGFR-TKI treatment (allowed treatment sequences: 1st+3rd generation, 2nd+3rd generation, or direct 3rd generation), no restriction on the number of prior chemotherapy lines, and stable parenchymal brain and extracranial lesions; ECOG Performance Status (PS) score of 0-3; normal major organ function, including hemoglobin (Hb) ≥90g/L, absolute neutrophil count (ANC) ≥1.5×10⁹/L, platelet (PLT) ≥100×10⁹/L, white blood cell count (WBC) ≥3.0×10⁹/L (without blood transfusion or hematopoietic stimulants within 14 days), alanine transaminase (ALT) and aspartate transaminase (AST) ≤2.5×upper limit of normal (ULN), total bilirubin (TBIL) ≤1.5×ULN, serum creatinine (Cr) ≤1.5×ULN or creatinine clearance ≥50ml/min (for patients with liver metastasis: TBIL ≤3×ULN, ALT and AST ≤5×ULN), activated partial thromboplastin time (APTT), international normalized ratio (INR), and prothrombin time (PT) ≤1.5×ULN, and left ventricular ejection fraction (LVEF) ≥50% by Doppler ultrasound; compliance with washout period requirements (≥21 days since the last chemotherapy dose if no prior radiotherapy, ≥14 days since the end of local radiotherapy for parenchymal brain metastases, ≥30 days since surgical resection of parenchymal brain metastases with full recovery from acute toxicity); expected survival time ≥3 months; ability to swallow oral medications (or receive crushed medications via gastrostomy tube if unable to swallow); for women of childbearing age, negative pregnancy test (serum or urine) within 14 days before enrollment and agreement to use effective contraception during the study and for 3 months after the last study drug administration; for men, surgical sterilization or agreement to use effective contraception during the same period; voluntary participation, signed informed consent (or by legal representative), and good expected compliance with study procedures.

   2.2 Exclusion Criteria Participants will be excluded if they meet any of the following: major surgery within 4 weeks before the start of study treatment or planned surgery during the study; human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS); active bacterial or fungal infections requiring intravenous antibiotics at the start of study treatment; history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid treatment, or signs of clinically active interstitial lung disease; arterial/venous thromboembolic events within 6 months before enrollment (including cerebrovascular accident, deep vein thrombosis, or pulmonary embolism); significant cardiovascular disease history (New York Heart Association class >2 congestive heart failure, unstable angina, myocardial infarction within 3 months before signing the informed consent form, symptomatic arrhythmias requiring treatment, or mean corrected QT interval (QTcF) >470ms on 3 consecutive electrocardiograms); history of other systemic malignant tumors within 5 years (excluding cured basal cell carcinoma of the skin, carcinoma in situ of the cervix, and ovarian cancer); use of drugs or supplements known to be strong inducers of CYP3A4; known allergy to any study drug or its excipients; pregnancy, lactation, or refusal of effective contraception by patients of childbearing potential; history of definite neurological or psychiatric disorders (including epilepsy and dementia); other conditions deemed unsuitable for enrollment by the investigator.
3. Study Design and Treatment Regimen 3.1 Study Design This is an open-label, single-arm Phase II prospective study with no randomization or blinding. The planned sample size is 30 patients, calculated based on a Pearson chi-square test to detect an increase in clinical response rate from 40% to 80% (power=0.8, one-sided significance level=0.20, 10% dropout rate).

   3.2 Treatment Regimen The combined treatment includes three components: double-dose third-generation EGFR-TKI (oral osimertinib 160mg once daily, furmonertinib 160mg once daily, or almonertinib 220mg once daily); intrathecal pemetrexed (administered via lumbar puncture, Ommaya reservoir, or intrathecal pump, with induction phase: 10mg twice weekly for 4 weeks, maintenance phase: 10mg once weekly for 4 weeks, consolidation phase: 30mg every 4 weeks until disease progression or intolerable toxicity); and bevacizumab 7.5mg/kg administered intravenously.

   3.3 Dose Adjustment and Management For missed doses: if vomiting occurs shortly after drug administration, no re-dose is given; for missed doses within 2 hours of the scheduled time, the dose is supplemented, otherwise, it is skipped without cycle adjustment. For intrathecal pemetrexed, administration requires ANC ≥1.5×10⁹/L, PLT ≥75×10⁹/L, Hb ≥80g/L, and ≤Grade 2 fatigue, oral mucositis, or neurotoxicity; for Grade ≥3 hematological or non-hematological toxicity, the next dose is reduced by 10mg. For bevacizumab, Grade 3-4 related adverse events (AEs) require treatment suspension until recovery to ≤Grade 1, then resumption at the original dose; permanent discontinuation is considered if toxicity fails to resolve or poses ongoing risks.
4. Study Procedures 4.1 Screening Period (D-28 to D-1) Within 28 days before enrollment, participants complete informed consent signing, collection of demographic and medical history data, tumor imaging (chest/abdominal/pelvic CT/MRI within 4 weeks), echocardiogram, drug allergy history review, and concurrent medication documentation. Within 14 days before drug administration, additional assessments include ECOG PS scoring, physical examination, laboratory tests (blood routine, urine routine, blood biochemistry, stool occult blood, coagulation function), electrocardiogram, pregnancy test, myocardial enzyme profile, HIV/hepatic B/hepatic C screening, thyroid function test, and CSF examination. Eligibility is confirmed only after all inclusion and exclusion criteria are met.

   4.2 Treatment Period In Cycle 1 (Month 1), assessments include vital signs, physical examination, AE monitoring, concurrent medication recording, and drug administration on Day 1; ECOG PS scoring, laboratory tests, electrocardiogram, and AE monitoring on Day 14; and imaging assessment on Day 28. For Cycle 3 and beyond, Day 1 assessments are the same as Day 14 of Cycle 1, Day 14 includes ECOG PS scoring, vital signs, physical examination, and AE monitoring, and imaging assessment is performed on Day 56. Imaging assessment frequency is every 4 weeks for the first 2 cycles, then every 8 weeks, and every 12 weeks after 1 year of follow-up. Extracranial lesions are evaluated per RECIST v1.1, and intracranial lesions per RANO-LM criteria.

   4.3 Follow-up Period Safety follow-up is conducted 30 days after the last study drug administration, repeating the assessments performed at treatment termination. Survival follow-up occurs every 3 months ±14 days to collect survival status and subsequent treatment information, with imaging assessments as per the treatment period schedule until new anticancer treatment initiation or disease progression.
5. Study Endpoints 5.1 Primary Endpoint The primary endpoint is leptomeningeal metastasis overall response rate (LM-ORR) evaluated by RANO-LM criteria.

   5.2 Secondary Endpoints Secondary endpoints include quality of life (QoL) assessed by the QLQ-C30 scale; leptomeningeal metastasis progression-free survival (LM-PFS), defined as the time from treatment initiation to LM progression or death; overall survival (OS), defined as the time from treatment initiation to death or last follow-up; improvement and duration of neurological symptoms/signs (from the date of significant/partial improvement to deterioration due to LM progression); improvement and duration of ECOG PS (from the date of ECOG score improvement to deterioration due to LM progression); and safety profile.

   5.3 Exploratory Endpoint The exploratory endpoint is the correlation between CSF genetic characteristics and prognosis/efficacy prediction in patients with LM following resistance to standard-dose third-generation EGFR-TKI.
6. Statistical Analysis Three analysis populations are defined: Full Analysis Set (all enrolled patients who received at least one dose of study drug), Per-Protocol Set (subset of Full Analysis Set without major protocol deviations), and Safety Analysis Set (all enrolled patients with at least one post-baseline safety assessment). Efficacy analysis uses the Kaplan-Meier method for survival curve estimation (OS, LM-PFS) and 95% confidence intervals, Fisher's exact test for comparing clinical response rates between subgroups, and Log-rank test for survival time comparisons. Statistical analyses are performed using SPSS 25.0 or Prism 8 software, with two-sided P<0.05 considered statistically significant.
7. Safety Evaluation AEs are collected from informed consent signing to 30 days after the last study drug administration, including onset time, severity (per NCI-CTCAE v5.0), duration, management, and outcome. Serious adverse events (SAEs) are defined as events leading to death, life-threatening conditions, hospitalization/prolonged hospitalization, permanent disability, congenital anomalies, or requiring medical intervention to prevent severe outcomes. SAEs must be reported to the ethics committee, NMPA, and relevant authorities within 24 hours of investigator awareness. For pregnant female participants, study drug is discontinued immediately, and follow-up continues until 1 month post-delivery; adverse pregnancy outcomes are reported as SAEs.
8. Data Management and Quality Assurance Case Report Forms (CRFs) are completed accurately and verified against original medical records, with all data modifications dated, signed, and explained without obscuring original entries. A dedicated data manager establishes and maintains the database, resolves data queries with investigators, and coordinates database locking with the principal investigator, statistician, and monitor. Data security is ensured through restricted access and regular backups, with any modifications requiring joint approval. Quality assurance measures include compliance with the Declaration of Helsinki (2008) and GCP guidelines, prior ethics committee approval of the study protocol and informed consent form, GCP training for study personnel, regular monitoring to ensure protocol adherence, and audits by regulatory authorities and the ethics committee.
9. Study Drugs Third-generation EGFR-TKIs include osimertinib (AstraZeneca, 80mg tablet, oral administration, sealed storage at ≤25℃), furmonertinib (Alivia, 40mg tablet, oral administration, sealed storage at ≤25℃), and almonertinib (Hansoh, 55mg tablet, oral administration, sealed storage at ≤25℃). Intrathecal pemetrexed (Qilu Pharmaceutical, 500mg lyophilized powder, intrathecal injection, sealed storage at 0-4℃) and bevacizumab (Qilu Pharmaceutical, 100mg:4ml injection, intravenous infusion, protected from light at 2-8℃, no freezing or vigorous shaking) are also used. All drugs are stored and administered per manufacturer's recommendations and study protocol requirements.

ELIGIBILITY:
Inclusion Criteria

* Aged ≥ 18 years at the time of signing the informed consent form, regardless of gender.
* Histologically or cytologically confirmed advanced or metastatic non-small cell lung cancer (NSCLC), staged as IV according to the 8th edition of the IASLC TNM classification (2015).
* Presence of EGFR-sensitive mutations (exon 19 deletion or exon 21 L858R mutation).
* Leptomeningeal metastasis (LM) progression after standard-dose first-, second-, or third-generation EGFR-TKI treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Adequate major organ function, defined as: hemoglobin (Hb) ≥ 90 g/L, absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L, platelet count (PLT) ≥ 100 × 10^9/L, white blood cell count (WBC) ≥ 3.0 × 10^9/L and ≤ 10.0 × 10^9/L; total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN), alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 2.5 × ULN; creatinine clearance ≥ 50 ml/min (for patients with liver metastases, TBIL ≤ 3.0 × ULN, ALT and AST ≤ 5.0 × ULN); activated partial thromboplastin time (APTT), international normalized ratio (INR), and prothrombin time (PT) ≤ 1.5 × ULN.
* At least 21 days since the last radiotherapy (including whole-brain radiotherapy or local radiotherapy for brain metastases).
* Expected survival ≥ 3 months.
* Ability to swallow oral medications (or receive crushed medications via gastrostomy tube if unable to swallow).
* For women: Agreement to use effective contraception (e.g., surgical sterilization or protocol contraception) within 14 days prior to enrollment, during the study, and for 3 months after the last study drug administration.
* For men: Agreement to use effective contraception (e.g., surgical sterilization or protocol contraception) during the study and for 3 months after the last study drug administration.
* Voluntary participation, signed informed consent, and willingness to comply with study procedures and protocols.

Exclusion Criteria

* Major surgery within 4 weeks prior to the start of study treatment, or need for major surgery during the study.
* Human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS).
* Active bacterial/fungal/viral infections requiring intravenous antibiotic therapy.
* Drug-induced pneumonitis or interstitial lung disease, or evidence of clinically significant active pulmonary disease.
* Severe cardiovascular events within 6 months prior to enrollment, including cerebrovascular accident, deep vein thrombosis, or pulmonary embolism.
* Significant cardiovascular disease, such as New York Heart Association (NYHA) class II or higher congestive heart failure, unstable angina, symptomatic arrhythmias requiring treatment, or corrected QT interval (QTcF) > 470 ms on consecutive electrocardiograms.
* History of other systemic malignant tumors within the past 5 years (except for cured basal cell carcinoma, carcinoma in situ of the cervix, and ovarian cancer).
* Use of drugs or supplements known to be strong inducers of CYP3A4.
* Known severe allergy to any study drug or its excipients.
* Pregnancy, lactation, or refusal of effective contraception by patients of childbearing potential.
* History of definite neurological or psychiatric disorders (including epilepsy and dementia).
* Other conditions deemed unsuitable for enrollment by the investigator.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
LM-ORR | Up to 30 days after the last study drug administration (for safety and response assessment), and through study completion, an average of 1 years (for survival follow-up)
  The primary endpoint is leptomeningeal metastasis overall response rate (LM-ORR) evaluated by RANO-LM criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No